CLINICAL TRIAL: NCT04506086
Title: A Phase 4, Multi-center Open-label Feasibility Study to Evaluate Outpatient Blinatumomab Administration in Adult Subjects With Minimal Residual Disease (MRD) of B-precursor Acute Lymphoblastic Leukemia (ALL) in Complete Hematologic Remission
Brief Title: Feasibility Study to Evaluate Outpatient Blinatumomab in Subjects With Minimal Residual Disease (MRD) of B-precursor Acute Lymphoblastic Leukemia (ALL)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The decision to terminate is not based on safety or efficacy but due to slow enrollment impacting the ability to complete the study as planned.
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20190014
Record Dates: First submitted 2020-07-27; First posted 2020-08-10 (Actual); Results first posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-04

CONDITIONS: B-precursor Acute Lymphoblastic Leukemia
Keywords: Blinatumomab; Leukemia; Acute lymphoblastic leukemia; B-precursor Acute Lymphoblastic Leukemia; Minimal/Measurable Residual Disease; Bi-specific T-cell engager
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Neoplasm, Residual | interventions — blinatumomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Blinatumomab (Experimental)
  Interventions: Drug: Blinatumomab; Device: Current Wearable Heatlth Monitoring System (CWHMS)

INTERVENTIONS:
Drug: Blinatumomab — Participants will receive blinatumomab continuous IV infusion for a maximum of 4 cycles. Each cycle is 6 weeks in duration consisting of 4 weeks of treatment and 2 weeks of rest.
  Other Names: AMG 103; Blincyto
Device: Current Wearable Heatlth Monitoring System (CWHMS) — The study will use the CWHMS device to monitor participants' vital signs while they are at home.

SUMMARY:
The study aims to determine the safety and feasibility of complete outpatient blinatumomab administration for subjects with minimal/measurable residual disease (MRD) of B-precursor Acute Lymphoblastic Leukemia (ALL).

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided informed consent prior to initiation of any study-specific activities/procedures OR subject's legally acceptable representative has provided informed consent prior to any study-specific activities/procedures being initiated when the subject has any kind of condition that, in the opinion of the Investigator, may compromise the ability of the subject to give written informed consent
* Age greater than or equal to 18 years
* B-cell precursor (BCP) acute lymphoblastic leukemia (ALL) with minimal/measurable residual disease defined as hematologic complete remission (CR) with less than 5% bone marrow blasts and meets clinical eligibility criteria to receive blinatumomab as outlined below.
* Hematologic criteria for remission as defined below:

  * Less than 5% bone marrow blasts
  * Absolute neutrophil count greater than or equal to 1.0 x10^9 L
  * Platelets greater than or equal to 50 x10^9/L (transfusion permitted)
  * Hemoglobin level greater than or equal to 90 g/L (transfusion permitted)
* Renal and hepatic function as defined below:
* Total bilirubin <3 x upper limit of normal (ULN) unless related to Gilbert's or Meulengracht disease
* Serum creatinine <1.5 x ULN. If serum creatinine ≥1.5 x ULN, then measure Glomerular Filtration Rate (GFR); subject will be eligible only if measured GFR is within normal limits.
* Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 or 1
* Negative pregnancy test in women of childbearing potential
* Ability and willingness to wear and comply with the instructions for the use of and monitoring of the digital monitoring devices as outlined in informed consent
* Subject resides within 1 hour of ground transportation to an advanced medical care facility for the duration of the mandatory device monitoring period (MDMP)
* Adequate cellular service available during MDMP.
* Presence of an adult (greater than or equal to 18 years) caregiver(s) in the same dwelling, for 24 hours/day for the entire MDMP. Caregiver will be expected to have access to transportation
* Ability and willingness to participate in the health management of the subject and to assist with the requirements of remote digital monitoring devices during the blinatumomab infusion within the MDMP

Exclusion Criteria:

* Presence of circulating blasts
* Presence of extramedullary disease
* History of relevant central nervous system (CNS) pathology or current relevant CNS pathology (seizure, paresis, aphasia, cerebrovascular ischemia/hemorrhage, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, psychosis, or coordination or movement disorders
* Current infiltration of cerebrospinal fluid (CSF) by ALL. If screening cerebrospinal fluid (CSF) demonstrates leukemic blasts, subjects must receive intrathecal treatment and demonstrate negative CSF before enrollment and starting blinatumomab infusion
* Current autoimmune disease or history of autoimmune disease with potential CNS involvement
* Allogeneic hematopoietic stem cell transplantation (HSCT) within 12 weeks before blinatumomab treatment
* Active acute or chronic graft versus host disease (GvHD) requiring systemic treatment with immunosuppressive medication
* Systemic chemotherapy within 2 weeks prior to study treatment (except for intrathecal prophylaxis)
* Radiotherapy within 4 weeks prior to study treatment
* Known hypersensitivity to blinatumomab or to any component of the product formulation
* Active malignancy other than ALL with the exception of basal cell or squamous cell carcinoma of the skin, or carcinoma in situ of the cervix
* History of other malignancy within the past 2 years, with the following exception[s]:

  * Malignancy treated with curative intent and with no known active disease present for greater than or equal to 2 years before enrollment and felt to be at low risk for recurrence by the treating physician
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated cervical carcinoma in situ without evidence of disease
  * Adequately treated breast ductal carcinoma in situ without evidence of disease
  * Prostatic intraepithelial neoplasia without evidence of prostate cancer
  * Adequately treated urothelial papillary non-invasive carcinoma or carcinoma in situ
* Currently receiving treatment with an investigational device or drug study or less than 30 days since ending treatment on an investigational device or drug study(ies)
* Active uncontrolled infection requiring therapy
* Known infection or chronic infection with hepatitis B virus (hepatitis B surface antigen [HBsAg] positive) or hepatitis C virus (HCV) (anti-HCV positive)
* Known positive test for human immunodeficiency virus (HIV)
* Any concurrent disease or medical condition deemed to interfere with the conduct of the study and remote digital monitoring as judged by the investigator
* Any acutely ill cardiac patients with the potential to develop life threatening arrhythmias eg, very fast atrial fibrillation
* Subjects with no cellular signal in their home
* Subjects with bi-lateral upper arm tattoos directly under the area of Current Wearable Health Monitoring System (CWHMS) application (Current Health wearable device)
* Subjects with a known allergy to any of the device component materials
* Subjects with open wounds on both arms directly under the area of CWHMS application (Current Health wearable device) or with injuries to both arms
* Subjects with an upper arm circumference of less than 20 cm or greater than 50 cm
* Subjects with an implantable defibrillator
* Subjects unwilling to wear the CWHMS (Current Health wearable device, axillary temperature patch) during the mandatory monitoring period (MDMP) in cycles 1 and 2
* Subjects with excessive scarring directly under the area of CWHMS (Current Health wearable device) application
* Subjects who cannot have their blood pressure (BP) measured in both arms (or wrists) eg due to atrio-venous shunt, risk of lymphedema or peripherally inserted central catheter line
* Female subject is pregnant or breastfeeding or planning to become pregnant or breastfeed during treatment and for an additional 48 hours after the last dose of protocol-specified therapy
* Female subjects of childbearing potential unwilling to use 1 highly effective method of contraception during treatment and for an additional 48 hours after the last dose of protocol-specified therapy Refer to Section 11.5 for additional contraceptive information
* Female subjects of childbearing potential with a positive pregnancy test assessed at Screening by a serum pregnancy test and/or urine pregnancy test
* Subject likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures (eg, patient reported outcomes [PROs]) to the best of the subject and investigator's knowledge

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-08-26 (Actual); Primary Completion 2024-07-04 (Actual); Study Completion 2024-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (12):
- United States (12):
  - City of Hope National Medical Center, Duarte, California
  - University of California Los Angeles, Los Angeles, California
  - University of California Irvine, Orange, California
  - Mayo Clinic, Jacksonville, Florida
  - Adventist Health System/Sunbelt, Inc d/b/a AdventHealth Orlando, Orlando, Florida
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Mount Sinai Hospital, New York, New York
  - University of Rochester Cancer Center, Rochester, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Saint Francis Hospital, Inc, Greenville, South Carolina
  - University of Virginia Health System, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 10 participants were enrolled in the United States from August 2021 to July 2024.
  This study was terminated by Amgen because of strategic reasons (slow enrollment) and not because of safety concerns.
Pre-assignment Details: Participants were administered blinatumomab as a continuous intravenous infusion (CiVI) in 2 mandatory cycles. Each cycle lasted 6 weeks (4 weeks of CiVI and 2-week treatment-free). Participants then had the option to continue for 2 additional cycles.
  Mandatory monitoring period (MDMP) was defined as the first 3 days of Cycle 1 and the first 2 days of Cycle 2.
  During MDMP, participants wore the current wearable health monitoring system to measure vital signs 24 hours a day.
Groups:
- Blinatumomab: Participants received 28 ug/day blinatumomab as a CiVI in two 6-week cycles.
Period: Overall Study
Arm/Group | Blinatumomab
Started | 10
Completed | 8
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: included all enrolled participants who receive at least 1 dose of blinatumomab.
Arm/Group | Blinatumomab
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 7
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Grade 3 and/or 4 Cytokine Release Syndrome (CRS), Neurotoxicity (NT) or Any Adverse Events Resulting in Hospitalization During MDMP
Description: Adverse event were graded using the Common Terminology Criteria for Adverse Events, (CTCAE) v5.0 grading Scale. Grade 3 events were defined as severe or medically significant but not immediately life-threatening; grade 4 events were defined as life-threatening consequences; urgent intervention indicated.
  CSR is a heightened T-cell activation and release of pro inflammatory cytokines. NT signs include encephalopathy, delirium, aphasia, lethargy, difficulty concentrating, agitation, tremor, seizures, and, rarely, cerebral edema.
Time Frame: Cycle 1: Day 1 to Day 3; Cycle 2: Day 1 and Day 2
Population: Safety Analysis Set included all enrolled participants who received at least 1 dose of blinatumomab.
Measure: Count of Participants; unit: Participants
Arm/Group | Blinatumomab
Number analyzed (Participants) | 10
Participants | 2

2. Secondary Outcome: Time to Therapeutic Intervention (TTI) During MDMP
Description: TTI was calculated for all the valid alarm triggers which lead to an intervention as duration (in minutes) from time of the device alert (alarm triggered) to the time of initiation of the therapeutic intervention.
  Therapeutic intervention was any measurable action taken by the participants or performed on the participants as a result of the onset of fever, hypotension, hypoxia, other grade 3 or 4 vital sign including seizure or neurological change (grade 3-limiting self-care activities of daily living [ADL]).
Time Frame: Cycle 1: Day 1 to Day 3; Cycle 2: Day 1 and Day 2
Population: Primary Analysis Set included all participants who received at least 1 dose of blinatumomab for whom the outpatient monitoring during blintumomab infusion was established.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Blinatumomab
Number analyzed (Participants) | 10
minutes | 14.98 (26.76)

3. Secondary Outcome: Number of Participants Experiencing Treatment-Emergent Adverse Events (TEAE) and Adverse Events of Interest (EOIs)
Description: TEAEs were defined as adverse events starting on or after first dose of blinatumomab. EOIs referred in particular to CRS, infections and neurologic events.
Time Frame: Up to a maximum of 193 days
Population: Safety Analysis Set included all enrolled participants who received at least 1 dose of blinatumomab.
Measure: Count of Participants; unit: Participants
Arm/Group | Blinatumomab
Number analyzed (Participants) | 10
Participants
  TEAEs | 10
  EOIs | 8

4. Secondary Outcome: Change From Baseline to Cycle 2 Day 1 in the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life of Cancer Patients (QLQ-C30) Global Health Status/ Quality of Life Score
Description: The EORTC QLQ-C30 is a 30-item questionnaire that assesses the health related quality of life of cancer patients participating in clinical trials. The EORTC QLQ-C30 forms a global health status (GHS)/quality of life (QoL) scale, 5 functional domains (physical, role, emotional, cognitive and social), and 9 symptom domains (fatigue, nausea and vomiting, pain, dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). All of the scales/items measures get mapped to a common range from 0 to 100. A high scale score represents a higher response level. Thus, a negative change for the global health status/QoL scale represents a lower QoL, a negative change for a functional scale represents a lower level of functioning, a positive change for a symptom scale/item represents a higher level of symptomatology/problems.
Time Frame: Baseline and Cycle 2 Day 1
Population: Patient-Reported Outcomes (PRO) Analysis Set included all participants in the safety analysis set with a non-missing baseline and at least 1 non-missing post-baseline result for EORTC QLQ-C30.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Blinatumomab
Number analyzed (Participants) | 4
score on a scale
  EORTC QLQ-C30 Global Health Status/QoL Score | -8.333 (11.785)
  EORTC QLQ-C30 Functional Scales Score | -12.778 (12.222)
  EORTC QLQ-C30 Symptoms Scales Score | 4.487 (6.743)

5. Secondary Outcome: Number of Participants Who Experienced TEAEs That Resulted in Hospitalization, Surgeries, Use of Concomitant Medications or Use of Device/Procedure Intervention
Description: Concomitant therapies are any concomitant medications or treatments deemed necessary to provide adequate supportive care except for:
  Any anti-tumor therapy other than the protocol-specified therapy (ie, radiation therapy, immunotherapy, cytotoxic and/or cytostatic drugs); Chronic systemic (> 7 days) high-dose corticosteroid therapy (dexamethasone > 24 mg/day or equivalent); any other immunosuppressive therapies (except for transient use of corticosteroids); Any other investigational agent. Intervention is any measurable action taken by the subject or performed on the subject as a result of the onset of a TEAE.
Time Frame: Up to a maximum of 193 days
Population: Safety Analysis Set included all enrolled participants who received at least 1 dose of blinatumomab.
Measure: Count of Participants; unit: Participants
Arm/Group | Blinatumomab
Number analyzed (Participants) | 10
Participants
  Hospitalizations | 3
  Surgeries | 0
  Use of concomitant medications | 9
  Use of device/procedure intervention | 3

ADVERSE EVENTS:
Time Frame: Up to a maximum of 193 days
Description: All-cause mortality is reported for all participants enrolled/randomized in the study. Serious adverse events and other adverse events are reported for all participants who received at least one dose of study drug.
Groups:
- Blinatumomab: Blinatumomab 28 ug/24h CIV open label
Arm/Group | Blinatumomab
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 4/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Blinatumomab (N=10)
Pyrexia (General disorders) | 1
Cytokine release syndrome (Immune system disorders) | 1
Sepsis (Infections and infestations) | 1
Encephalopathy (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Blinatumomab (N=10)
Neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Palpitations (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 2
Vision blurred (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Chills (General disorders) | 2
Fatigue (General disorders) | 2
Malaise (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 3
Cytokine release syndrome (Immune system disorders) | 3
Hypersensitivity (Immune system disorders) | 1
Candida infection (Infections and infestations) | 1
Enterocolitis infectious (Infections and infestations) | 1
Subcutaneous abscess (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Vascular access complication (Injury, poisoning and procedural complications) | 1
Blood creatinine increased (Investigations) | 1
Human rhinovirus test positive (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
White blood cell count decreased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 3
Tremor (Nervous system disorders) | 3
Confusional state (Psychiatric disorders) | 1
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 2
Superficial vein thrombosis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2022-04-21): https://cdn.clinicaltrials.gov/large-docs/86/NCT04506086/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-26): https://cdn.clinicaltrials.gov/large-docs/86/NCT04506086/SAP_001.pdf